CLINICAL TRIAL: NCT07008001
Title: Clinical Assessment of DOT Spectacle Lenses in Chinese Children Extension
Brief Title: Assessment of DOT Spectacles in Chinese Children Extension
Acronym: CATHAY Ext
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPRO-2201-002
Record Dates: First submitted 2025-05-14; First posted 2025-06-06 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Juvenile Myopia; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator/Investigational site staff tasked with measuring key primary variables (i.e., axial length and SER) will be masked to participant's former treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- SightGlass Vision Test Arm Groups I (formerly test group) (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Novel spectacle lens design
- SightGlass Vision Test Arm Groups II (formerly control group) (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Novel spectacle lens design

INTERVENTIONS:
Device: Novel spectacle lens design — Use of spectacle lenses may reduce the rate of progression of juvenile myopia

SUMMARY:
This is a randomized, controlled, open-label, evaluator-blinded, multicenter, clinical trial of 12-months duration to evaluate the continued safety and efficacy of Diffusion Optics Technology (DOT) spectacle lenses in reducing the progression of juvenile myopia in children of Chinese origin.

ELIGIBILITY:
Inclusion Criteria:

1. Previously a successfully completed participant in the CATHAY study (NCT05562622)
2. Agree to wear the assigned spectacles constantly except for sleeping, swimming, or other activities in which spectacle wear would be dangerous or otherwise not possible (minimum of 10 hours per day)
3. Willingness to participate in the trial for 12 months without contact lens wear or any other myopia management intervention
4. The subject's parent(s) or legal guardian(s) must read, understand and sign the Statement of Informed Consent and receive a fully executed copy of the form

Exclusion Criteria:

1. Known allergy to proparacaine, tetracaine, or tropicamide or cyclopentolate

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Axial length Group I | 12 months
  Change in axial length from baseline to 36 months
Axial length Group II | 12 months
  Change in axial length from baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Aier Eye Hospital, Changsha
  - West China Hospital, Chengdu
  - Zhongshan Ophthalmic Center, Guangzhou
  - Fudan University EENT, Shanghai
  - Tianjin Eye Hospital, Tianjin